CLINICAL TRIAL: NCT04395417
Title: Injection Therapy in Patients With Lateral Epicondylitis: Hyaluronic Acid or Prolotherapy?
Brief Title: Injection Therapy in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zilan Bazancir Apaydın, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/12
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: Lateral epicondylitis; Prolotherapy; Hyaluronic acid
MeSH Terms: conditions — Tennis Elbow | interventions — Hyaluronic Acid; Prolotherapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: The patients and the researcher who were responsible for the analyzing of the data were blinded to the randomization results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid injection group (Experimental): This is the study group in whom Hyaluronic acid injection was injected at lateral epicondylitis site.
  Interventions: Drug: Hyaluronic Acid
- Prolotherapy injection group (Active Comparator): This is the control group in whom prolotherapy injection was given at lateral epicondyle site.
  Interventions: Biological: Prolotherapy

INTERVENTIONS:
Drug: Hyaluronic Acid — Patients were infiltrated with injection single dose 30 mg/2 ml 1500 kilodalton high molecular weight hyaluronic acid at the lateral epicondyle according to the standard technique.
  Other Names: Prostrolane
  Arms: Hyaluronic acid injection group
Biological: Prolotherapy — Patients were infiltrated with 5cc of dextrose 15% at the lateral epicondyle according to the standard technique. For solution, 1 cc 2% lidocaine, 5 cc 30% hypertonic dextrose and 4 cc 0.9 % isotonic were used.
  Arms: Prolotherapy injection group

SUMMARY:
Lateral epicondylitis is a painful enthesopathy of the common extensor tendon at the lateral part of the elbow, with a prevalence of 1-3 % in the general population. In the treatment of lateral epicondylitis, the role of biological-based therapies has begun to investigate regeneration and optimize tendon healing. Prolotherapy (PrT) and hyaluronic acid (HA) injections are biological based treatments. Previous studies have shown benefit of PrT in the treatment of tendinopathies. Preliminary findings demonstrated that HA could be clinically effective in the treatment of enthesopathies. Considering the paucity of HA studies (which also lack a control group) and the proposed mechanism of action of both PrT and HA is through cell proliferation and the healing process of tendons, this study was conducted to compare the effect of PrT and HA in chronic lateral epicondylitis .

DETAILED DESCRIPTION:
Lateral epicondylitis and other chronic tendinopathies are now understood to be non-inflammatory conditions characterized by collagen degeneration, fibroblast proliferation, mucoid degeneration and neovascularization Biological-based treatments can trigger the release of cytokines and growth factors from platelets, leukocytes, macrophages and other inflammatory cells. These growth factors support neovascularization and the chemotaxis of fibroblasts and tenocytes. It stimulates proliferation and collagen remodeling of fibroblasts and tenocytes.

PrT involves multiple injections of a small amount of irritant or sclerosing solution. Common irritants include hypertonic dextrose, phenol-glycerin-glucose and sodium morrhuate. PrT injection mechanism is as follows; while hypertonic dextrose causes cell rupture through osmosis, monosodium morrhuate attracts inflammatory mediators and improves blood flow of the diseased tendon.Previous studies have shown benefit of PrT in the treatment of tendinopathies HA injection is a treatment method that increases the ability of sliding with its viscoelastic properties, reduces tendon surface friction and accelerates regeneration. In vitro models suggest that HA can increase collagen I production and accumulation with a dose-dependent positive collagen I / collagen III ratio. However, controlled randomised studies are still needed.

Mechanism of action of both PrT and HA is cell proliferation and the healing process of tendons, this study was conducted to compare the effect of PrT and HA in chronic lateral epicondylitis .

ELIGIBILITY:
Inclusion Criteria:

1. aged 20-60 years,
2. had a clinical diagnosis of lateral epicondylitis, defined as pain over the lateral humeral epicondyle of at least 6 months' duration,
3. provoked by palpation and resisted wrist/middle finger extension or gripping,
4. participants needed to score at least 30/100 on Visual analogue scale (VAS),
5. be able to understand enough Turkish to complete the outcome questionnaire.

Exclusion Criteria:

1. Any treatment for their elbow pain by a health care practitioner within the preceding 6 months,
2. Concomitant neck or other arm pain causing disability or requiring treatment within the last 6 months,
3. Clinical evidence of other primary sources of lateral elbow pain,
4. Upper limb fractures within the preceding 10 years,
5. Prior elbow surgery
6. Elbow steroid injection in the past 3 months
7. Systemic inflammatory disorder or malignancy,
8. Pregnancy or breastfeeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Pain via Visual Analogue Scale | Baseline, 6 week, 12 week
  Change from baseline at 6 week and at 12 week
  Pain of the participants will be assessed by most widely used and accepted "visual analogue scale". It consists of a 10 centimeter line marked at one end with "no pain" and at other end with "worst pain ever". Participant is asked to indicate where on the line he or she rates the pain on the day of presentation, baseline, 6 and 12 weeks of follow-ups. Numerical score is given to it simply by measuring length between "no pain" to patients mark.
Quick - Disabilities of the Arm, Shoulder and Hand (QuickDASH) | Baseline, 6 week, 12 week
  Change from baseline at 6 week and at 12 week
  The elbow disability scale was assessed using the Quick DASH (disability of arm, shoulder & hand) questionnaire containing 11 questions with five choices for each question. The final score can range between 0 (best condition) and 100 (worst condition). Participant is asked to answer the Quick DASH at baseline, 6 and 12 weeks of follow-ups

SECONDARY OUTCOMES:
Grip strength via dynamometer | Baseline, 6 week, 12 week
  Change from baseline at 6 week and at 12 week
  Pain-free grip strength is a commonly used objective measure of lateral epicondilitis-related disability with high reliability and validity. In the study, we used a hand dynamometer (Baseline® Hydraulic Hand Dynamometer 200 LB Standard). Patients were asked to sit, adduct the shoulder, flex the elbow to 90 degrees and put their forearm in a neutral position, then squeeze the dynamometer for three to five seconds. This test was conducted three times with 60-second intervals for each patient, and the mean patient grip strength was recorded at baseline, 6 and 12 weeks of follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal Altay, MD, Study Director — Inonu University Faculy of Medicine
Locations (1):
- Hakan Apaydın, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 12 months after publication
Access Criteria: Access criteria IPD and additional supporting information will share, analysis of primer and sekonder outcomes and clinical data will share after publication,

REFERENCES:
- [Derived] Apaydin H, Bazancir Z, Altay Z. Injection Therapy in Patients with Lateral Epicondylalgia: Hyaluronic Acid or Dextrose Prolotherapy? A Single-Blind, Randomized Clinical Trial. J Altern Complement Med. 2020 Dec;26(12):1169-1175. doi: 10.1089/acm.2020.0188. Epub 2020 Sep 15. PMID 32931308

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04395417/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04395417/ICF_001.pdf